CLINICAL TRIAL: NCT01758887
Title: Antipsychotic Discontinuation in High-risk Subjects
Status: Withdrawn | Type: Observational
Why Stopped: administrative reason
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jun Soo Kwon, Professor, Seoul National University Hospital
Other Study IDs: H-1207-055-417
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controls: Healthy control
- patients: clinical high risk subjects for psychosis

SUMMARY:
* Would be there any difference in dopamine synthesis between remitted clinical high risk subjects for psychosis and healthy control?
* What would happen to dopamine synthesis after antipsychotic discontinuation in clinical high risk subjects for psychosis?
* What about the dopamine synthesis in recurred clinical high risk subjects for psychosis after the discontinuation?

DETAILED DESCRIPTION:
After the antipsychotic medication discontinuation, we are going to assess the changes of the biological markers

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as a clinical High Risk
* Treated with antipsychotic drugs
* PSP1-5 (from SIPS criteria) <3 (severity index)for more than 6 months
* Had not experienced a symptomatic relapse in the 6 months

Exclusion Criteria:

* Significant abnormality in laboratory tests
* History of head trauma

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Clinical high risk subjects for psychosis who have been treated with antipsychotic medication so that reach to the remission.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Presynaptic dopamine synthesis in the striatum | baseline
  measured with [18F]DOPA positron emission tomography

CONTACTS AND LOCATIONS:
Overall Officials: Jun Soo Kwon, MD PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No